CLINICAL TRIAL: NCT02264795
Title: Does Intraperitoneal Instillation of Lidocaine at Cesarean Delivery Improve Postoperative Analgesia? A Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Does Intraperitoneal Instillation of Lidocaine at Cesarean Delivery Improve Postoperative Analgesia?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-04
Record Dates: First submitted 2014-10-09; First posted 2014-10-15 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Pain
Keywords: Cesarean section; Lidocaine
MeSH Terms: conditions — Pain | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Intraperitoneal instillation of normal saline.
  Interventions: Drug: Placebo
- Lidocaine (Active Comparator): Intraperitoneal instillation lidocaine 2% (400mg) with epinephrine 5mcg/ml.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Lidocaine 2% with epinephrine 5mcg/ml
  Other Names: Lidocaine HCl
  Arms: Lidocaine
Drug: Placebo — 0.9% Sodium Chloride Solution
  Other Names: Normal saline
  Arms: Placebo

SUMMARY:
The instillation of local anesthetic into the peritoneum has been found to be safe and effective in reducing postoperative pain and morphine consumption after abdominal surgery. A review of studies reporting serum levels of local anesthetic after intraperitoneal delivery found no cases of clinical toxicity in any of the trials. The studies in this meta-analysis did not include post-cesarean delivery pain and there is a lack of data to support the use of intraperitoneal local anesthetic after cesarean section.

The purpose of this study is to assess the efficacy of intraperitoneal lidocaine on postoperative pain scores after cesarean delivery. This study will compare a 20ml solution of lidocaine (400mg) with epinephrine 5mcg/ml versus normal saline (placebo) instilled into the peritoneum at the end of surgery in women undergoing cesarean delivery. The investigators hypothesize that intraperitoneal lidocaine will result in lower pain scores, reduce opioid consumption and opioid related side effects, and higher maternal satisfaction after cesarean delivery.

DETAILED DESCRIPTION:
Postoperative pain after cesarean delivery can have a significant negative impact on the mother's ability to care for her newborn and lead to complications such as thromboembolism, chronic pain, and depression. Postoperative analgesia for cesarean delivery has undergone remarkable improvement and is currently based on a multimodal approach to improve pain control and reduce the systemic complications of opiates. Despite this some patients still experience moderate to severe pain after cesarean delivery, and further strategies to improve analgesia and postoperative recovery are warranted.

The use of intraperitoneal local anesthetics to reduce postoperative pain has been studied in a variety of surgical settings, such as hysterectomy, laparoscopic cholecystectomy and minor laparoscopic gynecological procedures. These studies have compared different local anesthetics and the timing of local anesthetic delivery in relation to surgery, for example pre-procedure, at the end of surgery or via continuous catheter infusion. Intraperitoneal lidocaine at the end of surgery was associated with lower postoperative pain scores after total abdominal hysterectomy (200mg lidocaine) and laparoscopic cholecystectomy (400mg lidocaine). There is a large growing body of evidence to support the use of intraperitoneal local anesthetic to reduce postoperative pain. However, there is a lack of data to support its use in postcesarean delivery pain. The investigators found one study reporting a decreased incidence of postoperative pain following intraperitoneal lidocaine instillation at the end of cesarean delivery, in which the parietal peritoneum had been sutured.

The purpose of this study is to evaluate the efficacy of intraperitoneal lidocaine 400mg instillation at the end of cesarean delivery on maternal pain scores and satisfaction, in the context of a multimodal analgesic regimen inclusive of intrathecal opioids and systemic NSAIDs, acetaminophen and opioids. The investigators hypothesize that intraperitoneal lidocaine will decrease VAS pain scores, reduce opioid consumption and opioid related side effects, and increase maternal satisfaction after cesarean delivery.

ELIGIBILITY:
Inclusion Criteria:

* ASA I or II patients
* 18-50 years of age
* Term pregnancy
* Singleton pregnancy
* Spinal anesthetic
* Pfannenstiel incision
* Patients who have given pre-operative informed written consent

Exclusion Criteria:

* Patients who refuse or are unable to give consent
* ASA >2
* Multiple gestation
* Chronic pain
* BMI >40
* Contraindication to acetaminophen or non-steroidal anti-inflammatory drugs

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 204 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Pain Score (VAS) 24hr movement | 24 hours
  VAS score (VAS 0-100 mm) for maternal pain on movement at 24 hours postcesarean delivery

SECONDARY OUTCOMES:
Anxiety score before surgery (VAS) | 5 minutes
  Maternal anxiety score before surgery
Pain score (VAS) 2hr rest | 2 hours
  VAS score (VAS 0-100 mm) for maternal pain at rest at 2 hours postcesarean
Pain score (VAS) 2hr movement | 2 hours
  VAS score (VAS 0-100 mm) for maternal pain on movement at 2 hours postcesarean
Pain Score (VAS) 24hr rest | 24 hours
  VAS score (VAS 0-100 mm) for maternal pain at rest at 24 hours postcesarean
Pain Score (VAS) 48hr rest | 48 hours
  VAS score (VAS 0-100 mm) for maternal pain at rest at 48 hours postcesarean
Pain Score (VAS) 48hr movement | 48 hours
  VAS score (VAS 0-100 mm) for maternal pain on movement at 48 hours postcesarean
Patient satisfaction 2hr | 2 hours
  Patient satisfaction at 2 hours postcesarean
Patient satisfaction 24hr | 24 hours
  Patient satisfaction at 24 hours postcesarean
Patient satisfaction 48hr | 48 hours
  Patient satisfaction at 48 hours postcesarean
Opiate consumption PACU | 2 hours
  Opiate consumption on discharge from PACU
Opiate consumption 24hrs | 24 hours
  Opiate consumption within 24 hours postcesarean
Opiate consumption 48hrs | 48 hours
  Opiate consumption within 48 hours postcesarean
Side Effect scores | 48 hours
  Nausea, vomiting and pruritis scores on discharge from PACU, at 24 hours and 48 hours postcesarean
Bowel function | 48 hours
  Return of bowel function as assessed by passing flatus
Time to request for first opiate | 48 hours
  Hours to request for first opiate (if any) postcesarean

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Siddiqui, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada